CLINICAL TRIAL: NCT06672471
Title: Post-Operative Antibiotic Efficacy in Clean Contaminated Head and Neck Surgery: A Randomized Controlled Trial
Acronym: PEACH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Awais Kanwal, Dr. Muhammad Awais Kanwal Department of Surgical Oncology, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB-24-32
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Neoplasms; UADT Neoplasm; Cancer of the Head and Neck; Antibiotic Resistant Infection; Antibiotic Side Effect
Keywords: head; neck; cancer; surgery; ENT; Antibiotics
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: To determine whether postoperative antibiotic prophylaxis is necessary in patients undergoing Clean-contaminated head and neck surgery, or if a single perioperative antibiotic dose suffices.
  Primary Outcome Measure:
  Incidence of Surgical Site infection (SSI) This will be assessed on Post Operative Physical Clinic visits and will be recorded by an assessor who will be blind to whether the patient received Post Operative antibiotic or not.
  Secondary Outcome Measure:
  Post-Operative Complications The Secondary outcome measure, post-operative complications will be recorded as per the Clavien Dindo Classification (CDC)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study uses a triple blinded trial design to reduce bias, ensuring that neither the primary clinical teams, the patients, nor the post-operative assessors know the assigned treatment groups. The surgical and anesthetic teams performing the operation are blinded to group allocation, following standard care protocols without knowing if a patient receives postoperative antibiotics. Similarly, assessors who evaluate patients for surgical site infections (SSIs) during follow-up are blinded, preventing any influence on SSI assessment from knowledge of the patient's treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group Post operative Antibiotics (Active Comparator): A Single dose of Peri-Operative Antibiotic at the time of induction of Anaesthesia before incision for surgery is made and additional Post Operative Antibiotics for one day.
  Antibiotic to be used: Cefazolin 2 Gram IV Once followed by Cefazolin 1 Gram TID
  Interventions: Other: Post Operative Antibiotics for one day
- Intervention Group No Post Operative Antibiotics (Experimental): A Single dose of Peri-Operative Antibiotic at the time of induction of Anaesthesia before incision for surgery is made, the time of Antibiotics will be recorded in time-out form as a part of the surgical safety checklist.
  Antibiotic to be used: Cefazolin 2 Gram IV Once
  Interventions: Other: No Post Operative Antibiotics for intervention group

INTERVENTIONS:
Other: No Post Operative Antibiotics for intervention group — No Post Operative Antibiotics in patients going clean contaminated head and neck surgery
  Arms: Intervention Group No Post Operative Antibiotics
Other: Post Operative Antibiotics for one day — Control group will receive perioperative as well as post operative antibiotics for one day
  Arms: Control Group Post operative Antibiotics

SUMMARY:
The "Post-Operative Antibiotic Efficacy in Clean Contaminated Head and Neck Surgery" (PEACH) trial is a study designed to assess the necessity of post-operative antibiotics for preventing surgical site infections (SSIs) in clean-contaminated head and neck surgeries. Recognizing the pivotal role antibiotics have played since their discovery in reducing postoperative infections, this trial aims to determine if a single perioperative antibiotic dose can effectively prevent SSIs, or if additional post-operative antibiotics are required.

This study addresses a critical issue in the context of rising antibiotic resistance by potentially limiting unnecessary antibiotic use post-surgery while ensuring patient safety. Results could inform future guidelines, optimizing antibiotic use in surgical prophylaxis and contributing to global efforts against antibiotic resistance.

DETAILED DESCRIPTION:
In the pre-antibiotic era, surgery was a perilous endeavour, fraught with high infection risks and grim patient outcomes. Surgeons waged a relentless battle against postoperative infections. Even routine procedures were laden with danger, leading to severe complications, high morbidity, and alarming mortality rates. The inability to curb bacterial growth in surgical wounds cast a dark shadow over the medical field, highlighting the desperate need for a revolutionary breakthrough in infection control.

The Discovery of Penicillin in 1928 by Sir Alexander Fleming marked the beginning of the Antibiotic revolution On November 28, 1942, a fire broke out at The Cocoanut Grove Nightclub, in Boston, Massachusetts, and many survivors received skin grafts which are liable to infection by Staphylococcus. Treatment with penicillin was hugely successful at the Massachusetts General Hospital. Dozens of people were rescued from near-certain death in the first public demonstration of the powers of the antibiotic, at that time the Boston Globe called it "priceless" and Time magazine dubbed it a "wonder drug. This midwifed the birth of the modern pharmaceutical industry, and nearly doubled life expectancy, from 48 years at the turn of the 20th century to 78 years in the post-World War II years.

This also provided hope for surgeons grappling with the scourge of Surgical Site Infections. Antibiotics emerged as powerful weapons in the arsenal against infectious complications, ushering in a new era of proactive infection control. For the first time, surgeons had tools to combat bacteria directly, significantly reducing postoperative complications. This newfound ability to administer antibiotics prophylactically before surgical incisions marked a profound turning point, ultimately enhancing patient safety and reshaping the surgery landscape.

Despite the remarkable achievements, the euphoria surrounding antibiotics precipitated a darker issue. The widespread and indiscriminate administration of antibiotics, sometimes in situations where they confer minimal benefit, sowed the seeds of a formidable adversary: Antibiotic Resistance. The emergence of antibiotic-resistant strains of bacteria represents an enduring challenge in modern healthcare. The overreliance on these powerful drugs inadvertently fostered the survival of resistant organisms, diminishing the effectiveness of antibiotics over time. This challenge reverberates across various medical contexts, including surgical prophylaxis, reminding us of the importance of judicious antibiotic use.

The threat of antibiotic resistance is real. Therefore, all the stakeholders must employ strategies to prevent and control antibiotic resistance to prevent an imminent post-antibiotic era, a condition that may be worse than the pre-antibiotic era.

Resistant organisms are difficult to treat, requiring higher doses or alternative drugs, which are possibly more toxic and expensive. According to the Centre for Disease Control and Prevention (CDC), at least 2 million people become infected with antibiotic-resistant bacteria and more than 23,000 people die annually as a consequence of these infections. This is expected to be more in developing countries where communicable diseases remain the leading causes of death. To worsen the situation are the emerging and re-emerging infectious diseases, lack of development of new classes of antibiotics and continuing increasing antibiotic resistance, including superbugs (bacteria with accumulated resistance to almost all available antibiotics), at alarming and dangerous levels worldwide.

In the current state of the field of antimicrobials, resistance is certainly not limited to clinical microbiology as it was in the early years of the antibiotic era. Thus, it is not a single grand challenge; it is rather a complex problem requiring the concerted efforts of microbiologists, ecologists, health care specialists, educationalists, policymakers, legislative bodies, agricultural and pharmaceutical industry workers, and the public to deal with.

This should be of everyone's concern, because, in the end, there is always a probability for any of us at some stage to get infected with a pathogen that is resistant to antibiotic treatment. Moreover, even behavioural patterns, such as hygienic habits or compliance with antibiotic treatment regimens, may have consequences that are not limited only to individual health issues but, on a larger scale, contribute to antibiotic resistance.

In an era of increasing antibiotic resistance, maintaining a delicate balance between effective prophylaxis and judicious antibiotic use is paramount. [9]. The Centres for Disease Control and Prevention (CDC) divides surgical wounds into four categories: clean, clean-contaminated, contaminated, and dirty operative wounds. In head and neck surgery, many procedures are clean, i.e., creating wounds without contact with the upper aerodigestive tract (UADT) (e.g., thyroidectomy). In this group, SSIs occur in less than 1% .

Major procedures with exposure to the UADT (e.g., Partial Glossectomy, Buccal mucosal resection and reconstructions, laryngectomy) are considered "clean-contaminated". The UADT harbours a large variety of microorganisms, such as gram-positive and facultative anaerobic bacteria, and to a lesser degree gram-negative bacteria, Candida species, and bacteria originating from an eventually harvested flap.

Surgeons, infection control specialists, and researchers must unite to enhance current protocols and investigate innovative approaches to ensure patient safety during surgical procedures. This study aims to determine if a single perioperative dose of antibiotics is sufficient to reduce surgical site infections (SSIs) in clean-contaminated head and neck surgeries or if postoperative antibiotic administration is necessary.

By pursuing this research, The Investigators envision a future where our collective efforts control antimicrobial resistance, make SSIs a rare occurrence rather than a common risk, and significantly improve the quality of surgical care and patient outcomes.

This study will be conducted as a double-blinded trial, ensuring that neither the primary clinical teams nor the patients are aware of the assigned treatment group, which minimizes bias and enhances the objectivity of the results.

The surgical and anaesthetic teams, responsible for performing and managing the operation, will be blinded to the group allocation. They will not have access to the randomization assignments and will treat all patients as per standard care without knowledge of whether postoperative antibiotics are being administered. The team evaluating patients for surgical site infections (SSIs) in the post-operative follow-up clinic will also be blinded. These assessors will not know whether patients belong to the intervention or control group, which prevents any influence on SSI assessment based on knowledge of the patient's post operative antibiotic treatment.

The assignment to either the intervention or control group will be randomized and kept confidential. Only essential personnel, such as a Nurse, pharmacist or designated study member will access the randomization information to dispense the appropriate treatment (antibiotics or placebo) as per the protocol. This data will not be shared with the surgical, anaesthetic, or postoperative assessment teams.

To ensure patient blinding, those in the control group will receive a placebo identical in appearance to the antibiotic prescribed to the intervention group. The patients will not be informed of whether they are receiving active antibiotics or a placebo postoperatively, reducing the risk of patient behavior or reporting being influenced by their treatment group.

In the intervention group, patients will receive perioperative antibiotics only, administered during the induction of anesthesia, before the surgical incision is made, with no postoperative antibiotics given. In contrast, the control group patients will be given antibiotics postoperatively for one day, simulating standard practice. The patient's medication will be indistinguishable from the placebo given to the intervention group, ensuring they are unaware of their group allocation.

Through these blinding measures, the study aims to reduce potential biases in treatment administration, SSI assessment, and patient-reported outcomes. This rigorous blinding design will contribute to the reliability and validity of the study's findings on the effectiveness of perioperative-only versus extended postoperative antibiotic prophylaxis.

Pre-operative randomization after enrolment will be carried out and patients will be allocated either to the "intervention group" or to the "Control group" by "computerized block randomization". Research Randomizer software, a free-to-use software will be used for this. Patients will be randomized either into the intervention group or into the control group.

Patients will be enrolled pre-operatively, in clinics while booking for surgery. The researcher responsible for enrolment will ensure that the patient understands the study completely and can comprehend his/her role.

The researcher will inform the enrolled patients about the randomization and will tell them that the enrolled patients will have equal chances of ending up in the "Intervention group" or the "Control" and the enrolled patients must not share the details of medication received to the assessor as it may lead to a bias, contact details of Primary investigator will be shared with the enrolled patients to ensure that all their queries and concerns are addressed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and older.
2. Patients undergoing elective Clean-contaminated head and neck surgery.
3. Patients who have provided informed consent.
4. Patients with a life expectancy of more than 6 months.

Exclusion Criteria:

1. Patients aged less than 18.
2. Patients with a history of antibiotic allergies.
3. Patients with ongoing infections or those requiring preoperative antibiotics.
4. Patients with immunocompromised conditions (e.g., HIV, on immunosuppressive therapy).
5. Patients undergoing emergency surgery.
6. Patients undergoing palliative surgery.
7. Patients undergoing Clean Head and Neck Surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical Site Infection | 4 weeks after surgery
  This will be assessed on Post Operative Physical Clinic visits and will be recorded by an assessor who will be blind to whether the patient received Post Operative antibiotic or not. SSI will be determined using a Clinical Examination and the findings will be recorded, pictures of the wound will be taken at every visit for up to four weeks to be uploaded in the patient's electronic records to be viewed later, A Standardized assessment (Looking for Spreading erythema, Localised pain, Pus or discharge from the wound, Persistent pyrexia, wound dehiscence) will be carried out by the clinician and the findings will be documented in patient electronic records in hospital information system (HIS).

SECONDARY OUTCOMES:
Rate of Post Operative Complications | 4 weeks after surgery
  The Secondary outcome measure, post-operative complications will be recorded as per the Clavien Dindo Classification (CDC)
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusions and total parenteral nutrition are also included. Grade III Requiring surgical, endoscopic or radiological intervention Grade III a Intervention not under general anaesthesia Grade III b Intervention under general anaesthesia Grade IV Life-threatening complications (including CNS complications) * (requiring ICU management) Grade IV a single organ dysfunction (including dialysis) Grade IV b Multi-organ Dysfunction Grade V Death of a patient

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Syed Raza Hussain Consultant Oro-Maxillo-Facial Surgeon, MBBS, BDS, FDSRCS (ENG,IRL), Study Chair — Shaukat Khanum Memorial Cancer Hospital and Research Centre; Dr. Muhammad Faisal Consultant Head & Neck Surgery, BDS,FCPS,FHNS, Study Chair — Shaukat Khanum Memorial Cancer Hospital and Research Centre; Dr. Shayan Khalid Ghaloo Senior Instructor Head & Neck Surg., MBBS,FCPS, Study Director — Shaukat Khanum Memorial Cancer Hospital and Research Centre; Dr. Muhammad Awais Kanwal, MBBS,B.Sc, Principal Investigator — Shaukat Khanum Memorial Cancer Hospital and Research Centre
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital and Research Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Yes, we plan to share Individual Participant Data (IPD) that is non-identifiable. This data will be available once the study is completed and the results have been published. Individual requests can be directed to Dr. Muhammad Awais Kanwal at awaiskanwal@gmail.com or Dr. Shayan Khalid Ghaloo at shayankhalid@skm.org.pk.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We Plan to Share once study has been concluded.
Access Criteria: Requests will be seen on case to case basis.

REFERENCES:
- [Background] Watson AP, Tullo AB, Kerr-Muir MG, Ridgway AE, Lucas DR. Arborescent bacterial keratopathy (infectious crystalline keratopathy). Eye (Lond). 1988;2 ( Pt 5):517-22. doi: 10.1038/eye.1988.101. PMID 3256489
- [Background] Righi M, Manfredi R, Farneti G, Pasquini E, Cenacchi V. Short-term versus long-term antimicrobial prophylaxis in oncologic head and neck surgery. Head Neck. 1996 Sep-Oct;18(5):399-404. doi: 10.1002/(SICI)1097-0347(199609/10)18:53.0.CO;2-0. PMID 8864730
- [Background] Koshkareva YA, Johnson JT. What is the perioperative antibiotic prophylaxis in adult oncologic head and neck surgery? Laryngoscope. 2014 May;124(5):1055-6. doi: 10.1002/lary.24226. Epub 2013 Jun 10. No abstract available. PMID 23754680
- [Background] Dhole S, Mahakalkar C, Kshirsagar S, Bhargava A. Antibiotic Prophylaxis in Surgery: Current Insights and Future Directions for Surgical Site Infection Prevention. Cureus. 2023 Oct 28;15(10):e47858. doi: 10.7759/cureus.47858. eCollection 2023 Oct. PMID 38021553
- [Background] Shlykov IP. [Effect of somatotropin on the thyroid gland regeneration in hypophysectomized rats]. Probl Endokrinol (Mosk). 1969 Sep-Oct;15(5):69-74. No abstract available. Russian. PMID 5354621
- [Background] Alanis AJ. Resistance to antibiotics: are we in the post-antibiotic era? Arch Med Res. 2005 Nov-Dec;36(6):697-705. doi: 10.1016/j.arcmed.2005.06.009. PMID 16216651
- [Background] Adedeji WA. THE TREASURE CALLED ANTIBIOTICS. Ann Ib Postgrad Med. 2016 Dec;14(2):56-57. No abstract available. PMID 28337088
- [Background] Stewart CL. The fire at Cocoanut Grove. J Burn Care Res. 2015 Jan-Feb;36(1):232-5. doi: 10.1097/BCR.0000000000000111. PMID 25094013
- [Background] Fleming A. On the antibacterial action of cultures of a penicillium, with special reference to their use in the isolation of B. influenzae. 1929. Bull World Health Organ. 2001;79(8):780-90. No abstract available. PMID 11545337
- [Background] Aminov RI. A brief history of the antibiotic era: lessons learned and challenges for the future. Front Microbiol. 2010 Dec 8;1:134. doi: 10.3389/fmicb.2010.00134. eCollection 2010. PMID 21687759